CLINICAL TRIAL: NCT05562076
Title: A Prospective, Multicenter, Randomized Controlled Trail Using Spot Stenting to Treat Lower Extremity Post-angioplasty Dissection
Brief Title: Clinical Study of Focal Implant Used for Lower Extremity Post-angioplasty Dissection
Acronym: PINTO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhejiang Zylox Medical Device Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 72202207
Record Dates: First submitted 2022-08-15; First posted 2022-09-30 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Peripheral Artery Disease
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Drug Delivery Systems

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ZENFLEX ® Pinto (Experimental): subjects using the spot stent(ZENFLEX ® Pinto) system
  Interventions: Device: the spot stent(ZENFLEX ® Pinto) system
- Everflex (Active Comparator): subjects using the bare stent(Everflex) system
  Interventions: Device: the bare stent( Everflex) system

INTERVENTIONS:
Device: the spot stent(ZENFLEX ® Pinto) system — the spot stent(ZENFLEX ® Pinto) system、Color Doppler Ultrasonography (CDU) imaging、Dual Fluoroscopic Imaging、Digital subtraction angiography（DSA）
  Arms: ZENFLEX ® Pinto
Device: the bare stent( Everflex) system — the bare stent( Everflex) system、Color Doppler Ultrasonography (CDU) imaging、Dual Fluoroscopic Imaging、Digital subtraction angiography（DSA）
  Arms: Everflex

SUMMARY:
This is a prospective, multicenter, randomized controlled trail using spot stenting to treat lower extremity post-angioplasty dissection.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 80 years,male or female
2. Lower extremity atherosclerotic occlusive disease
3. After PTA, angiography showed less than 30% residual stenosis of the target lesion (based on visual estimation), and there is one or more dissection(Type A-F)
4. Subjects are able to understand the purpose of the study, demonstrate full compliance with the procedure and follow-up and sign informed consent

Exclusion Criteria:

1. The target lesion has been stented or previously treated with bypass surgery
2. Acute thrombosis of the target vessel requires thrombolysis or thrombectomy, or has undergone local or systemic thrombolysis within 48 hours
3. Cutting balloon, thrombectomy, plaque resection, brachytherapy, and laser therapy were planned
4. More than 30% residual stenosis of the inflow artery (based on visual estimation) after treatment, or there is no outflow artery in the target limb
5. The target lesion was too calcified to undergo PTA or the guide wire could not pass anterograde through the target lesion
6. Planned amputation on the target limb
7. Severe allergy to anticoagulant drugs, antiplatelet drugs, contrast media and Nitinol
8. Uncontrollable infections
9. Women who are pregnant or breastfeeding, or who plan to become pregnant during the duration of the trial
10. Participating in clinical trials of any other drug or medical device and not yet out of the study
11. Other circumstances not suitable for inclusion as judged by the investigator

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 224 (Estimated)
Dates: Start 2022-11 (Estimated); Primary Completion 2024-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
primary patency rate at 12 months after operation | 12 months

SECONDARY OUTCOMES:
success rate of the device | Intraoperation
success rate of the technique | post operation
rate of CD-TLR | 6 months,12 months
ABI | post operation, 6 months,12 months
Rutherford classification | post operation, 6 months,12 months
the incidence of major adverse events | 30 days, 6 months,12 months
the rate of target limb major amputation | 30 days, 6 months,12 months
the incidence of adverse events | Intraoperation, post operation, 30 days, 6 months,12 months
the incidence of SAE | Intraoperation, post operation, 30 days, 6 months,12 months
the rate of device defect | Intraoperation, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoqiang Li, Principal Investigator — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Locations (12):
- China (12):
  - Xuanwu Hospital, Capital Medical University, Beijing
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu
  - Changzhou First People's Hospital, Changzhou
  - Changzhou Second People's Hospital, Changzhou
  - The First Affiliated Hospital of Harbin Medical University, Ha’erbin
  - Anhui Provincial Hospital, Hefei
  - The Second Affiliated Hospital of Nanchang University, Nanchang
  - Nanjing Drum Tower Hospital, Nanjing
  - Affiliated Hospital of Qingdao University, Qingdao
  - Shanghai Ninth People's Hospital, Shanghai
  - Tianjin Medical University General Hospital, Tianjin
  - North Jiangsu People's Hospital, Yangzhou